CLINICAL TRIAL: NCT00472082
Title: An Open Label, Single-Center Pilot Study of Early Conversion From Tacrolimus to Efalizumab Maintenance Therapy in Primary Renal Transplant Recipients
Brief Title: Early Conversion From Tacrolimus to Efalizumab Maintenance Therapy in Kidney Transplant Recipients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated at the request of the drug manufacturer.
Sponsor: Emory University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Kenneth Newell, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003005; ACD4056s (Other: Other)
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2012-12-06 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Transplantation; Chronic Kidney Failure
Keywords: Immunosuppression; Renal Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): The study drug Efalizumab will be given as part of a triple drug regimen including mycophenolate mofetil and prednisone. A test dose of Efalizumab 0.7mg/kg will be given at the enrollment visit. Beginning with study visit 2, Efalizumab 1mg/kg will be administered subcutaneously by injection on a weekly basis for 1 year. Mycophenolate mofetil will be given at a dose of 2gm/day which is the same as the standard of care dose. If patient experiences drug toxicity with mycophenolate mofetil they may be reduced and resume a minimum of at least 1gram daily to continue in the study. Patients will be maintained at 10mg of prednisone daily, same as standard of care.
  Interventions: Drug: efalizumab

INTERVENTIONS:
Drug: efalizumab — Administration of a test dose of efalizumab 0.7mg/kg will be administered at enrollment. Weekly subcutaneous injections of efalizumab 1mg/kg will begin with study visit 2 and continue for 1 year for this pilot study.
  Other Names: Raptiva is the brand name FDA approved for the treatment of psoriasis.

SUMMARY:
The toxicity of calcineurin inhibitors(CNI)is a major factor limiting the success of renal transplantation. This protocol aims to replace the calcineurin inhibitor, tacrolimus, with efalizumab early after transplantation in patients with mild impairment of renal function in order to minimize the toxicities of CNI.

DETAILED DESCRIPTION:
Over the last two decades there have been significant improvements in renal transplantation due in large part to the decreasing incidence of acute rejection (down to less than 20% for first renal transplants) with the use of calcineurin inhibitors (CNI) such as cyclosporin and tacrolimus. Though proven very effective anti-rejection medications their use is associated with adverse side effects, including high blood pressure, post transplant diabetes, and high cholesterol, predisposing risk factors for cardiovascular disease and cerebrovascular disease. Chronic use of these drugs has also waged limitations to the long term survival of transplanted kidneys and kidney recipients with an increase in the development of chronic allograft nephropathy (CAN). There is also an increased incidence of chronic renal failure in non renal transplant recipients receiving CNI based treatments.

The mechanism of action for these reagents is known to be imprecise and science has sought to replace the current therapies in place with less toxic drugs more specific in their signaling pathway targets. In recent years cell surface proteins, restricted to cells of the immune system have been identified as mediators of the rejection response. The activation of T cells has been seen to activate an immune response correlated clinically with rejection. Integrins, specifically leukocyte function associated antigen LFA-1, are cell surface molecules which play a role in T-cell activation. LFA-1 is made up of two subunits, known as CD11 and CD18. Efalizumab is a humanized monoclonal antibody against the CD11 molecule. By binding to CD11 on T cells the system blocks the interaction between LFA-1 and ICAM-1, an intercellular adhesion molecule also necessary for T cell activation, thereby diminishing an immune response. The blockade formed does not deplete the T cells.

There have been preliminary studies using efalizumab in combination with cyclosporine. A very low incidence of rejection was observed in all groups receiving efalizumab (7.8%). However 3 cases of post-transplant lymphoproliferative disease were seen in 38 patients. There have been no cases of lymphomas or lymphoproliferative disease reported in clinical trials evaluating efalizumab for the treatment of psoriasis, suggesting that the combination of efalizumab and cyclosporine may have resulted in over immunosuppression.

As per standard of care, recipients of a kidney transplant at Emory are managed with a combination of the calcineurin inhibitor Prograf (tacrolimus), Cellcept (an antiproliferative agent) and Prednisone, a corticosteroid. For this study the investigators have chosen to substitute efalizumab in place of Prograf, after 3 months post transplant the period where the incidence of acute rejection is highest. Efalizumab, known by its trade name Raptiva, was approved by the FDA in October 2003 for the treatment of psoriasis. It is hypothesized that the conversion from Prograf to efalizumab will be associated with improved renal function and not associated with an increased risk of rejection. The investigators hope to address the challenges faced by recipients of transplanted kidneys in the long course of their transplanted organ's management with more favorable alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Primary renal transplant recipients
* recipients of deceased donor or living donor transplant
* Age 18-65 years (inclusive)
* Male or female
* Within 3-9 month window post-transplantation
* No episodes of acute rejection prior to enrollment
* Mild impairment of renal function as defined by a calculated CrCl of 35-50 ml/min/m2

Exclusion Criteria:

* Subjects with any prior solid organ transplant (including kidney)
* Subjects with a history of panel-reactive antibodies greater than 20% or the development of new anti-HLA antibodies after transplantation and prior to enrollment
* Subjects the Investigator deems to be at a relatively higher risk for acute rejection
* HLA-identical living donor pairs
* Evidence of infection with Hepatitis C (antibody positive or PCR positive), Hepatitis B ( surface antigen positive), HIV
* Subjects with BK or CMV viremia prior to enrollment
* Multiple organ transplant recipients
* Subjects with underlying renal disease of focal segmental glomerulosclerosis, membranoproliferative glomerulonephritis, hemolytic-uremic syndrome/thrombocytopenic purpura syndrome (due to risk of rapid disease recurrence in the allograft
* EBV negative recipients
* Women who are pregnant or nursing
* Women of child bearing age unwilling or unable to use an acceptable method to avoid pregnancy for the duration of the study and up to 8 weeks after last injection
* Patients not able to tolerate a dose of at least 500 mg of mycophenolate mofetil twice daily
* Allergy to Iodine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Newell, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from population of stable renal transplant recipients being followed at the Emory Transplant Center
Groups:
- Efalizumab Conversion: The study drug Efalizumab will be given as part of a triple drug regimen including mycophenolate mofetil and prednisone. A test dose of Efalizumab 0.7mg/kg will be given at the enrollment visit. Beginning with study visit 2, Efalizumab 1mg/kg will be administered subcutaneously by injection on a weekly basis for 1 year. Mycophenolate mofetil will be given at a dose of 2gm/day which is the same as the standard of care dose. If patient experiences drug toxicity with mycophenolate mofetil they may be reduced and resume a minimum of at least 1gram daily to continue in the study. Patients will be maintained at 10mg of prednisone daily, same as standard of care.
  efalizumab : Administration of a test dose of efalizumab 0.7mg/kg will be administered at enrollment. Weekly subcutaneous injections of efalizumab 1mg/kg will begin with study visit 2 and continue for 1 year for this pilot study.
Period: Overall Study
Arm/Group | Efalizumab Conversion
Started | 5
Completed | 0
Not Completed | 5
Not completed — Study prematurely terminated | 5

BASELINE CHARACTERISTICS:
Arm/Group | Efalizumab Conversion
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Will be Determined by Change in Renal Function as Measured by Cold Iothalamate Glomerular Filtration Rate(GFR)3 Months After Enrollment, and Acute Rejection Episodes Within the First 6 Months Post Enrollment.
Time Frame: 6 months from conversion
Arm/Group | Efalizumab Conversion
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety, Including Incidence of Post- Transplant Infections, Malignancies, Morbidities, Hypertension, Glucose Intolerance, Serum Cholesterol and Triglycerides Profile Over Time, Development of New Anti-donor Antibodies.
Time Frame: 1 year
Arm/Group | Efalizumab Conversion
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs were collected on subjects from time of enrollment through early termination of the study in 02/2009
Arm/Group | Efalizumab Conversion
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Efalizumab Conversion (N=5)
Hospitalization (Infections and infestations) | 2/2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No